CLINICAL TRIAL: NCT01963429
Title: A Randomized Phase III Study of the Comparison Between Radiofrequency Ablation and Hypofractionated Proton Beam Radiation in Patients With Recurrent/Residual Small Hepatocellular Carcinoma (APROH Study)
Brief Title: Comparison Between Radiofrequency Ablation and Hypofractionated Proton Beam Radiation for Recurrent/Residual HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Joong-Won Park, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS 13-695
Record Dates: First submitted 2013-10-13; First posted 2013-10-16 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Recurrent Small Hepatocellular Carcinoma; Residual Small Hepatocellular Carcinoma
Keywords: hepatocellular; Proton; RFA
MeSH Terms: interventions — Radiofrequency Ablation; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A(radiofrequency ablation ) (Experimental): radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation
- B(Proton) (Experimental): hypofractionated proton beam therapy
  Interventions: Radiation: Proton beam therapy

INTERVENTIONS:
Procedure: radiofrequency ablation — * RFA(radiofrequency ablation )
  * RFA electrode: Cool-tip RF ablation system (Covidien plc, 20 Lower Hatch Street Dublin 2, Ireland) and Well-Point RF Electrode (STARmed, Koea)
  * performed using either the manufacturer's standard algorithm or an interactive algorithm, with the latter being used when the impedance did not begin to increase at the midinterval of the standard algorithm
  * the duration of a single RFA session was 10 min to 15 min.
  Arms: A(radiofrequency ablation )
Radiation: Proton beam therapy — * Proton
  66 GyE /10 fx, 6.6 GyE fraction dose, 5 days/week, for HCC free from the alimentary tract (i.e., stomach, duodenum, esophagus, small and large bowel) (more than 2cm from clinical target volume),TLV30<40%,and/orRLV30<30%)
  Arms: B(Proton)

SUMMARY:
This phase 3 study is to evaluate the effectiveness of the comparison between radiofrequency ablation and hypofractionated proton beam radiation.

DETAILED DESCRIPTION:
The sample size for this study was based on a non-inferiority design. Primary objective: estimate local progression-free survival (LPFS) rate in two treatments Primary endpoint: 2-year LPFS rate Expected 2-year LPFS rate in the RFA: 85% Accural time and follow up time: 24 months and 24 months, respectively. Precision for 2-year LPFS rate estimation: Allowing a difference of 15% as the non-inferiority margin, with a power of 80% and a type I error level of 5%, evaluable 68 patients are required.

Considering 5% of follow-up loss, we need 72 patients in each arm, so a total of 144 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed as (i) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level greater than 200 IU/ml and a radiologically compatible feature with HCC in one or more CT/MRI/angiograms, or (ii) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level less than 200 IU/ml, and a radiologically compatible feature with HCC in two or more CT/MRI/angiograms or (iii) histological confirmation
* HCC patients who had recurrent or residual tumor after other treatments
* without evidence of extrahepatic metastasis
* the largest diameter of tumor should be less than 3cm, and the number of tumor ≤2
* no previous treatment to target tumors by other forms of RT
* liver function of Child-Pugh class A or B7 (Child-Pugh score of ≤7)
* Age of ≥18 years
* performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score
* WBC count ≥ 2,000/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 50,000/mm3; and adequate hepatic function (total bilirubin ≤ 3.0 mg/dL; AST and ALT < 5.0× upper limit of normal; no ascites)
* no serious comorbidities other than liver cirrhosis
* written informed consent

Exclusion Criteria:

* evidence of extrahepatic metastasis
* age < 18 years
* liver function of Child-Pugh class B8-9 and C (Child-Pugh score of >7) or uncontrolled cases of active chronic hepatitis B
* previous history of other forms of RT adjacent to target tumors
* poor performance status of 3 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* pregnant or breast feeding status
* previous history uncontrolled other malignancies within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
local progression-free survival(LPES) | up to 2 year
  To evaluate the local progression-free survival for 2 years

SECONDARY OUTCOMES:
disease-free survival (DFS) | up to 2 years until study closed
  Disease-free survival was defined as the interval from the date of randomization to date of detection study closed

OTHER OUTCOMES:
overall survival (OS) | up to 2 years until study closed
  Overall survival(OS) was defined as the interval from the date of randomization to date of detection study closed

CONTACTS AND LOCATIONS:
Overall Officials: Joong Won Park, Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim TH, Koh YH, Kim BH, Kim MJ, Lee JH, Park B, Park JW. Proton beam radiotherapy vs. radiofrequency ablation for recurrent hepatocellular carcinoma: A randomized phase III trial. J Hepatol. 2021 Mar;74(3):603-612. doi: 10.1016/j.jhep.2020.09.026. Epub 2020 Oct 5. PMID 33031846